CLINICAL TRIAL: NCT04097483
Title: The TELE-DD Project: a Nurse-led Randomised Controlled Trial on Treatment Adherence in Patients With Type 2 Diabetes and Comorbid Depression
Brief Title: Treatment Adherence Intervention in Patients With Type 2 Diabetes and Comorbid Depression
Acronym: TELE-DD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alicia Monreal Bartolomé (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor-Investigator, Alicia Monreal Bartolomé, MS, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TELE-DD
Record Dates: First submitted 2019-09-16; First posted 2019-09-20 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2; Depression
Keywords: Comorbidity; Depression; Type 2 Diabetes; Primary Health Care; Randomized-Controlled Trial; Treatment Adherence; Telephone-Based Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Primary Care specialist will be blind, but the telephonic intervention research nurses will not. For ethical and practical reasons, the trial will be unmasked, and participants will not be blind to the treatment condition once allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Intervention Group (Experimental): Nurse-led, telephone-based, and psychoeducational intervention, centered on motivational interviewing and cognitive behavioural therapy for adherence and depression.
  Interventions: Behavioral: Telephone Intervention Group
- Control group (No Intervention): Control group with treatment as usual (TAU).

INTERVENTIONS:
Behavioral: Telephone Intervention Group — Nurse-led, telephone-based, and psychoeducational intervention centered on motivational interviewing and cognitive behavioral therapy for adherence and depression.
  Arms: Telephone Intervention Group

SUMMARY:
Patients with diabetes have higher depression rates, impaired QOL and increased mortality rates due to complications and comorbid depression. Nurse-led, telephonic-based, and psychoeducational interventions have separately proved to improve disease prognosis and emotional distress in diabetes, but no study has integrated previous research findings with collaborative care and strong methods centred in treatment adherence outcomes. The Telephonic Monitoring on Diabetes and co-morbid Depression (TELE-DD) Project includes a three-phased population-based cohort study and nurse-led randomised controlled trial. The proposed intervention, based on monthly structured telephone calls, unifies proved techniques like motivational interviewing, cognitive behavioural therapy and patient's healthy behaviours education.

The integration in the TELE-DD Project of previous clinical research and a robust epidemiological dual design, will improve treatment adherence and further prognosis in patients with type 2 diabetes and comorbid depression through maximising clinical outcomes improvement, while guaranteeing cost-effectiveness and the long-term sustainability of findings translation to PC clinical practice services and public health programs.

DETAILED DESCRIPTION:
Patients with diabetes mellitus have a depression rate 1.6-2 times higher, impaired quality of life and increased mortality rates due to complications, comorbid depression or both. Prognosis in diabetes and depression comorbidity can be improved by increasing treatment adherence. Nurse-led, telephonic-based, and psychoeducational interventions, centred on motivational interviewing and cognitive behavioural therapy for adherence and depression, have separately improved prognosis and emotional distress in diabetic patients with comorbid depression.

The Telephonic Monitoring on Diabetes and co-morbid Depression (TELE-DD) Project aims to integrate prior well-stablished clinical research with collaborative care. A whole population cohort of adults (21+) with type 2 diabetes (T2D) and comorbid depression from twenty-three Health Centres from a whole Health System Region in Spain, will be approached for inclusion in the TELE-DD Project (N=7,271). Patients with confirmed diagnoses and pharmacological treatment for both diseases will be included in Phase I baseline cohort. In Phase II, 400 participants diagnosed with depression and T2D with no treatment adherence will be selected to participate in the randomised controlled trial (RCT). The TELE-DD Project is a three-stage both observational and comparative effectiveness study that includes a population-based cohort study (Phases I and III), and a nurse-led randomised controlled trial (Phase II), aimed to compare a telephonic-based psychoeducational intervention (TIG) vs treatment as usual (TAU) to improve treatment adherence (TA), and a further two- to five-year prognosis and cost-effectiveness study, in T2D patients with comorbid clinical depression from Primary Care (PC) services.

The integration in the TELE-DD Project of previous clinical research and a robust epidemiological design, will improve treatment adherence and further prognosis in these through maximising clinical outcomes improvement, while guaranteeing cost-effectiveness and the long-term sustainability of findings translation to PC clinical practice services and public health programs.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (21+).
* Concurrent type 2 diabetes (T2D) and depression diagnose registered in the SALUD clinical computerised system before January 1st, 2016.
* A duration of both T2D and depression of at least one year.
* Willingness to follow the TELE-DD research nurse instructions including self-monitoring of blood glucose.
* Fluent in the Spanish language
* Provision of signed and dated informed consent prior to any study procedures.
* No treatment adherence to both T2D and depression, or treatment adherence to both.

Exclusion Criteria:

* Presence of hearing problems, Alzheimer Disease, dementia or another serious cognitive or psychiatric disorder.
* Use of private health insurance that may influence the RCT intervention outcomes.
* Absence of pharmacological treatment for T2D or depression according to the CHS-EMR.
* Change of address or place of residence out of SALUD Zaragoza Region II, or no access to a phone.
* No Primary Care Specialist (PCS) or inability to identify a reference one.
* Treatment adherence only for one of the two conditions (D2T or depression).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Diabetes control measured by Glycosylated Haemoglobin | Baseline
  In the Intervention and control group
Diabetes control measured by Glycosylated Haemoglobin | 6-month follow-up
  In the Intervention and control group
Diabetes control measured by Glycosylated Haemoglobin | 12-month follow-up
  In the Intervention and Control group
Diabetes control measured by Glycosylated Haemoglobin | 18-month follow-up
  In the Intervention and Control group
Patient Health Questionnaire (PHQ-9) | Baseline
  In the Intervention and Control group. The Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | 6-month follow-up
  In the Intervention and Control group. The Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | 12-month follow-up
  In the Intervention and Control group. The Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | 18-month follow-up
  In the Intervention and Control group. The Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Medication possession ratio (MPR) | Baseline
  In the Intervention and Control group. Medication adherence was assessed using the medication possession ratio (MPR). It is calculated as the proportion of the number of days with treatment provided during the intended period of treatment, that is, 100 × (days supplied) / 365. Once TA is computed, a dichotomous variable is created as TA (Yes/No) considering a cut-off ratio of MPR ≥80%.
Medication possession ratio (MPR) | 6-month follow-up
  In the Intervention and Control group. Medication adherence was assessed using the medication possession ratio (MPR). It is calculated as the proportion of the number of days with treatment provided during the intended period of treatment, that is, 100 × (days supplied) / 365. Once TA is computed, a dichotomous variable is created as TA (Yes/No) considering a cut-off ratio of MPR ≥80%.
Medication possession ratio (MPR) | 12-month follow-up
  In the Intervention and Control group. Medication adherence was assessed using the medication possession ratio (MPR). It is calculated as the proportion of the number of days with treatment provided during the intended period of treatment, that is, 100 × (days supplied) / 365. Once TA is computed, a dichotomous variable is created as TA (Yes/No) considering a cut-off ratio of MPR ≥80%.
Medication possession ratio (MPR) | 18-month follow-up
  In the Intervention and Control group. Medication adherence was assessed using the medication possession ratio (MPR). It is calculated as the proportion of the number of days with treatment provided during the intended period of treatment, that is, 100 × (days supplied) / 365. Once TA is computed, a dichotomous variable is created as TA (Yes/No) considering a cut-off ratio of MPR ≥80%.
MBG questionnaire | Baseline
  In the Intervention and Control group. The MBG questionnaire includes TA questions related to timely drug intake, diet, PCS visits, physical activity, self-management, and others; prior research showed a Cronbach's alpha of 69% and a total explained variance of 63%.
MBG questionnaire | 6-month follow-up
  In the Intervention and Control group. The MBG questionnaire includes TA questions related to timely drug intake, diet, PCS visits, physical activity, self-management, and others; prior research showed a Cronbach's alpha of 69% and a total explained variance of 63%.
MBG questionnaire | 12-month follow-up
  In the Intervention and Control group. The MBG questionnaire includes TA questions related to timely drug intake, diet, PCS visits, physical activity, self-management, and others; prior research showed a Cronbach's alpha of 69% and a total explained variance of 63%.
MBG questionnaire | 18-month follow-up
  In the Intervention and Control group. The MBG questionnaire includes TA questions related to timely drug intake, diet, PCS visits, physical activity, self-management, and others; prior research showed a Cronbach's alpha of 69% and a total explained variance of 63%.
LDL-Cholesterol | Baseline
  In the Intervention and Control group. LDL-C values were registered according to reference values and recommendations from the National Cholesterol Education Program Adult Treatment Panel III (2001): <100 mg/dl optimum, 100-129 mg normal or close to optimal level, 130-159 mg/dl normal-high, 160-189 mg/dl high,> 190 mg/dl very high.
LDL-Cholesterol | 6-month follow-up
  In the Intervention and Control group. LDL-C values were registered according to reference values and recommendations from the National Cholesterol Education Program Adult Treatment Panel III (2001): <100 mg/dl optimum, 100-129 mg normal or close to optimal level, 130-159 mg/dl normal-high, 160-189 mg/dl high,> 190 mg/dl very high.
LDL-Cholesterol | 12-month follow-up
  In the Intervention and Control group. LDL-C values were registered according to reference values and recommendations from the National Cholesterol Education Program Adult Treatment Panel III (2001): <100 mg/dl optimum, 100-129 mg normal or close to optimal level, 130-159 mg/dl normal-high, 160-189 mg/dl high,> 190 mg/dl very high.
LDL-Cholesterol | 18-month follow-up
  In the Intervention and Control group. LDL-C values were registered according to reference values and recommendations from the National Cholesterol Education Program Adult Treatment Panel III (2001): <100 mg/dl optimum, 100-129 mg normal or close to optimal level, 130-159 mg/dl normal-high, 160-189 mg/dl high,> 190 mg/dl very high.
Diabetes Distress Scale (DDS) | Baseline
  In the Intervention and Control group. Four main domains can be identified in DDS: emotional burden, physician-related distress, regimen-related distress, and interpersonal distress, as well as obtaining a total score. Previous analyses identified that DDS had good sensitivity (95%) and specificity (85%), and was considered a reliable (α = 0.93) instrument for clinical practice and research (Polonsky et al., 2005), and has been validated in Spanish language (Ortiz et al., 2013).
Diabetes Distress Scale (DDS) | 6-month follow-up
  In the Intervention and Control group. Four main domains can be identified in DDS: emotional burden, physician-related distress, regimen-related distress, and interpersonal distress, as well as obtaining a total score. Previous analyses identified that DDS had good sensitivity (95%) and specificity (85%), and was considered a reliable (α = 0.93) instrument for clinical practice and research (Polonsky et al., 2005), and has been validated in Spanish language (Ortiz et al., 2013).
Diabetes Distress Scale (DDS) | 12-month follow-up
  In the Intervention and Control group. Four main domains can be identified in DDS: emotional burden, physician-related distress, regimen-related distress, and interpersonal distress, as well as obtaining a total score. Previous analyses identified that DDS had good sensitivity (95%) and specificity (85%), and was considered a reliable (α = 0.93) instrument for clinical practice and research (Polonsky et al., 2005), and has been validated in Spanish language (Ortiz et al., 2013).
Diabetes Distress Scale (DDS) | 18-month follow-up
  In the Intervention and Control group. Four main domains can be identified in DDS: emotional burden, physician-related distress, regimen-related distress, and interpersonal distress, as well as obtaining a total score. Previous analyses identified that DDS had good sensitivity (95%) and specificity (85%), and was considered a reliable (α = 0.93) instrument for clinical practice and research (Polonsky et al., 2005), and has been validated in Spanish language (Ortiz et al., 2013).

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the Intervention group and the Control group
Blood pressure | Baseline
  Blood pressure was measured according to the Spanish Heart Society (Moliner de la Puente et al., 2008), which is based on the National Institute for Health and Clinical Excellence guidelines (NICE, 2011).
Blood pressure | 6-month follow-up
  Blood pressure was measured according to the Spanish Heart Society (Moliner de la Puente et al., 2008), which is based on the National Institute for Health and Clinical Excellence guidelines (NICE, 2011).
Blood pressure | 12-month follow-up
  Blood pressure was measured according to the Spanish Heart Society (Moliner de la Puente et al., 2008), which is based on the National Institute for Health and Clinical Excellence guidelines (NICE, 2011).
Blood pressure | 18-month follow-up
  Blood pressure was measured according to the Spanish Heart Society (Moliner de la Puente et al., 2008), which is based on the National Institute for Health and Clinical Excellence guidelines (NICE, 2011).
Body mass index (BMI) | Baseline
  Body mass index (BMI) calculated as weight in kilograms divided by height height in square meters. In patients who are overweight or obese, a moderate reduction in body weight (5-10% of weight) is associated with improved insulin sensitivity, better glycemic control, reduced triglycerides and increased serum c-HDL.
Body mass index (BMI) | 6-month follow-up
  Body mass index (BMI) calculated as weight in kilograms divided by height height in square meters. In patients who are overweight or obese, a moderate reduction in body weight (5-10% of weight) is associated with improved insulin sensitivity, better glycemic control, reduced triglycerides and increased serum c-HDL.
Body mass index (BMI) | 12-month follow-up
  Body mass index (BMI) calculated as weight in kilograms divided by height height in square meters. In patients who are overweight or obese, a moderate reduction in body weight (5-10% of weight) is associated with improved insulin sensitivity, better glycemic control, reduced triglycerides and increased serum c-HDL.
Body mass index (BMI) | 18-month follow-up
  Body mass index (BMI) calculated as weight in kilograms divided by height height in square meters. In patients who are overweight or obese, a moderate reduction in body weight (5-10% of weight) is associated with improved insulin sensitivity, better glycemic control, reduced triglycerides and increased serum c-HDL.
Research nurse qualitative and quantitative evaluation about Treatment Adherence and diseases management. | Baseline
  The research nurse will record her qualitative and quantitative evaluation on how she thinks the patient is responding to treatment adherence and any detail of both diabetes and depression management. This evaluation will include a quantitative measure containing a 1-5 scale and a qualitative recording. This assessment will serve as a reference to compare with the patients' responses.
Research nurse qualitative and quantitative evaluation about Treatment Adherence and diseases management. | 6-month follow-up
  The research nurse will record her qualitative and quantitative evaluation on how she thinks the patient is responding to treatment adherence and any detail of both diabetes and depression management. This evaluation will include a quantitative measure containing a 1-5 scale and a qualitative recording. This assessment will serve as a reference to compare with the patients' responses.
Research nurse qualitative and quantitative evaluation about Treatment Adherence and diseases management. | 12-month follow-up
  The research nurse will record her qualitative and quantitative evaluation on how she thinks the patient is responding to treatment adherence and any detail of both diabetes and depression management. This evaluation will include a quantitative measure containing a 1-5 scale and a qualitative recording. This assessment will serve as a reference to compare with the patients' responses.
Research nurse qualitative and quantitative evaluation about Treatment Adherence and diseases management. | 18-month follow-up
  The research nurse will record her qualitative and quantitative evaluation on how she thinks the patient is responding to treatment adherence and any detail of both diabetes and depression management. This evaluation will include a quantitative measure containing a 1-5 scale and a qualitative recording. This assessment will serve as a reference to compare with the patients' responses.

CONTACTS AND LOCATIONS:
Overall Officials: María-Luisa Lozano-del-Hoyo, MSc, Principal Investigator — Universidad de Zaragoza; María-Teresa Fernández-Rodrigo, PhD, Principal Investigator — Universidad de Zaragoza; Juan F Roy, PhD, Principal Investigator — Camilo Jose Cela University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agámez Paternina, A.P., Hernández Riera, R., Cervera Estrada, L., Rodríguez García, Y., 2008. Factores relacionados con la no adherencia al tratamiento antihipertensivo. Revista Archivo Médico de Camagüey, 12(5). ISSN 1025-0255.
- [Background] Aikens JE, Piette JD. Diabetic patients' medication underuse, illness outcomes, and beliefs about antihyperglycemic and antihypertensive treatments. Diabetes Care. 2009 Jan;32(1):19-24. doi: 10.2337/dc08-1533. Epub 2008 Oct 13. PMID 18852334
- [Background] Alam R, Sturt J, Lall R, Winkley K. An updated meta-analysis to assess the effectiveness of psychological interventions delivered by psychological specialists and generalist clinicians on glycaemic control and on psychological status. Patient Educ Couns. 2009 Apr;75(1):25-36. doi: 10.1016/j.pec.2008.08.026. Epub 2008 Dec 11. PMID 19084368
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] Alexander GC, Sehgal NL, Moloney RM, Stafford RS. National trends in treatment of type 2 diabetes mellitus, 1994-2007. Arch Intern Med. 2008 Oct 27;168(19):2088-94. doi: 10.1001/archinte.168.19.2088. PMID 18955637
- [Background] Al-Hayek AA, Robert AA, Alzaid AA, Nusair HM, Zbaidi NS, Al-Eithan MH, Sam AE. Association between diabetes self-care, medication adherence, anxiety, depression, and glycemic control in type 2 diabetes. Saudi Med J. 2012 Jun;33(6):681-3. No abstract available. PMID 22729127
- [Background] Ali S, Stone M, Skinner TC, Robertson N, Davies M, Khunti K. The association between depression and health-related quality of life in people with type 2 diabetes: a systematic literature review. Diabetes Metab Res Rev. 2010 Feb;26(2):75-89. doi: 10.1002/dmrr.1065. PMID 20186998
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2015. Diabetes Care 2015;38(Suppl. 1), S1-S94. https://doi.org/10.2337/diaclin.33.2.97
- [Background] Anderson RJ, Freedland KE, Clouse RE, Lustman PJ. The prevalence of comorbid depression in adults with diabetes: a meta-analysis. Diabetes Care. 2001 Jun;24(6):1069-78. doi: 10.2337/diacare.24.6.1069. PMID 11375373
- [Background] Andrade SE, Kahler KH, Frech F, Chan KA. Methods for evaluation of medication adherence and persistence using automated databases. Pharmacoepidemiol Drug Saf. 2006 Aug;15(8):565-74; discussion 575-7. doi: 10.1002/pds.1230. PMID 16514590
- [Background] Asche C, LaFleur J, Conner C. A review of diabetes treatment adherence and the association with clinical and economic outcomes. Clin Ther. 2011 Jan;33(1):74-109. doi: 10.1016/j.clinthera.2011.01.019. PMID 21397776
- [Background] Baader, M., Tomas, Molina, F., José Luis, Venezian, B., Silvia, Rojas, C., Carmen, Farías, S., Renata, Fierro-Freixenet, Carlos, Backenstrass, Mathias, Mundt, Christoph., 2012. Validación y utilidad de la encuesta PHQ-9 (Patient Health Questionnaire) en el diagnóstico de depresión en pacientes usuarios de atención primaria en Chile. Rev. Chil. de neuro-psiquiatr. 50(1), 10-22. https://dx.doi.org/10.4067/S0717-92272012000100002
- [Background] Campayo A, de Jonge P, Roy JF, Saz P, de la Camara C, Quintanilla MA, Marcos G, Santabarbara J, Lobo A; ZARADEMP Project. Depressive disorder and incident diabetes mellitus: the effect of characteristics of depression. Am J Psychiatry. 2010 May;167(5):580-8. doi: 10.1176/appi.ajp.2009.09010038. Epub 2010 Feb 1. PMID 20123914
- [Background] Catapano AL, Reiner Z, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman M, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; European Society of Cardiology (ESC); European Atherosclerosis Society (EAS). ESC/EAS Guidelines for the management of dyslipidaemias The Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Atherosclerosis. 2011 Jul;217(1):3-46. doi: 10.1016/j.atherosclerosis.2011.06.028. No abstract available. PMID 21882396
- [Background] Chireh B, D'Arcy C. Shared and unique risk factors for depression and diabetes mellitus in a longitudinal study, implications for prevention: an analysis of a longitudinal population sample aged ⩾45 years. Ther Adv Endocrinol Metab. 2019 Jul 25;10:2042018819865828. doi: 10.1177/2042018819865828. eCollection 2019. PMID 31384422
- [Background] De-la-Camara, C.; Gracia-Garcia, P.; Roy, J. F.; et al, 2010. Influence of gender on baseline characteristics of depression and future risk for incident stroke an elderly population: Results from the ZARADEMP project. Journal of Psychosomatic Research, 68(6), 618-618. Web of Science (WOS): 000278468200047. HTTPS://DOI.ORG/10.1111/cns.12339
- [Background] de Jonge P, Roy JF, Saz P, Marcos G, Lobo A; ZARADEMP Investigators. Prevalent and incident depression in community-dwelling elderly persons with diabetes mellitus: results from the ZARADEMP project. Diabetologia. 2006 Nov;49(11):2627-33. doi: 10.1007/s00125-006-0442-x. Epub 2006 Sep 21. PMID 17019601
- [Background] Delahanty LM, Grant RW, Wittenberg E, Bosch JL, Wexler DJ, Cagliero E, Meigs JB. Association of diabetes-related emotional distress with diabetes treatment in primary care patients with Type 2 diabetes. Diabet Med. 2007 Jan;24(1):48-54. doi: 10.1111/j.1464-5491.2007.02028.x. PMID 17227324
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] Egede LE, Nietert PJ, Zheng D. Depression and all-cause and coronary heart disease mortality among adults with and without diabetes. Diabetes Care. 2005 Jun;28(6):1339-45. doi: 10.2337/diacare.28.6.1339. PMID 15920049
- [Background] Fisher L, Glasgow RE, Strycker LA. The relationship between diabetes distress and clinical depression with glycemic control among patients with type 2 diabetes. Diabetes Care. 2010 May;33(5):1034-6. doi: 10.2337/dc09-2175. Epub 2010 Feb 11. PMID 20150291
- [Background] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Background] Fisher L, Mullan JT, Arean P, Glasgow RE, Hessler D, Masharani U. Diabetes distress but not clinical depression or depressive symptoms is associated with glycemic control in both cross-sectional and longitudinal analyses. Diabetes Care. 2010 Jan;33(1):23-8. doi: 10.2337/dc09-1238. Epub 2009 Oct 16. PMID 19837786
- [Background] Gonzalez JS, Peyrot M, McCarl LA, Collins EM, Serpa L, Mimiaga MJ, Safren SA. Depression and diabetes treatment nonadherence: a meta-analysis. Diabetes Care. 2008 Dec;31(12):2398-403. doi: 10.2337/dc08-1341. PMID 19033420
- [Background] Gonzalez JS, Tanenbaum ML, Commissariat PV. Psychosocial factors in medication adherence and diabetes self-management: Implications for research and practice. Am Psychol. 2016 Oct;71(7):539-551. doi: 10.1037/a0040388. PMID 27690483
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Grossman A, Grossman E. Blood pressure control in type 2 diabetic patients. Cardiovasc Diabetol. 2017 Jan 6;16(1):3. doi: 10.1186/s12933-016-0485-3. PMID 28056987
- [Background] Expert Dyslipidemia Panel; Grundy SM. An International Atherosclerosis Society Position Paper: global recommendations for the management of dyslipidemia. J Clin Lipidol. 2013 Nov-Dec;7(6):561-5. doi: 10.1016/j.jacl.2013.10.001. Epub 2013 Oct 22. PMID 24314355
- [Background] Haynes RB. Determinants of compliance: The disease and the mechanics of treatment. Compliance in health care. Baltimore, MD, Johns Hopkins University Press, 1979. https://doi.org/10.1016/S0197-0070(84)80012-1
- [Background] Hoogendoorn CJ, Roy JF, Gonzalez JS. Shared Dysregulation of Homeostatic Brain-Body Pathways in Depression and Type 2 Diabetes. Curr Diab Rep. 2017 Aug 16;17(10):90. doi: 10.1007/s11892-017-0923-y. PMID 28815394
- [Background] Hoogendoorn CJ, Shapira A, Roy JF, Walker EA, Cohen HW, Gonzalez JS. Depressive symptom dimensions and medication non-adherence in suboptimally controlled type 2 diabetes. J Diabetes Complications. 2019 Mar;33(3):217-222. doi: 10.1016/j.jdiacomp.2018.12.001. Epub 2018 Dec 7. PMID 30598369
- [Background] Ho PM, Rumsfeld JS, Masoudi FA, McClure DL, Plomondon ME, Steiner JF, Magid DJ. Effect of medication nonadherence on hospitalization and mortality among patients with diabetes mellitus. Arch Intern Med. 2006 Sep 25;166(17):1836-41. doi: 10.1001/archinte.166.17.1836. PMID 17000939
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; ISPOR Health Economic Evaluation Publication Guidelines-CHEERS Good Reporting Practices Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS)--explanation and elaboration: a report of the ISPOR Health Economic Evaluation Publication Guidelines Good Reporting Practices Task Force. Value Health. 2013 Mar-Apr;16(2):231-50. doi: 10.1016/j.jval.2013.02.002. PMID 23538175
- [Background] Hutter N, Schnurr A, Baumeister H. Healthcare costs in patients with diabetes mellitus and comorbid mental disorders--a systematic review. Diabetologia. 2010 Dec;53(12):2470-9. doi: 10.1007/s00125-010-1873-y. Epub 2010 Aug 11. PMID 20700575
- [Background] International Diabetes Federation, 2017. IDF Diabetes Atlas (8th edition). International Diabetes Federation. https://www.idf.org/e-library/epidemiology-research/diabetes-atlas.html (accessed 20 April 2019).
- [Background] Ismail K, Winkley K, Rabe-Hesketh S. Systematic review and meta-analysis of randomised controlled trials of psychological interventions to improve glycaemic control in patients with type 2 diabetes. Lancet. 2004 May 15;363(9421):1589-97. doi: 10.1016/S0140-6736(04)16202-8. PMID 15145632
- [Background] Iverson, C., Christiansen, S., Flanigan, A., et al., 2007. AMA Manual of Style. 10th ed. New York, Oxford University Press, pp. 416-417.
- [Background] Johnson JA, Al Sayah F, Wozniak L, Rees S, Soprovich A, Chik CL, Chue P, Florence P, Jacquier J, Lysak P, Opgenorth A, Katon WJ, Majumdar SR. Controlled trial of a collaborative primary care team model for patients with diabetes and depression: rationale and design for a comprehensive evaluation. BMC Health Serv Res. 2012 Aug 16;12:258. doi: 10.1186/1472-6963-12-258. PMID 22897901
- [Background] Kreider KE. Diabetes Distress or Major Depressive Disorder? A Practical Approach to Diagnosing and Treating Psychological Comorbidities of Diabetes. Diabetes Ther. 2017 Feb;8(1):1-7. doi: 10.1007/s13300-017-0231-1. Epub 2017 Feb 3. PMID 28160185
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lee YJ, Kang HM, Kim NK, Yang JY, Noh JH, Ko KS, Rhee BD, Kim DJ. Factors associated for mild cognitive impairment in older korean adults with type 2 diabetes mellitus. Diabetes Metab J. 2014 Apr;38(2):150-7. doi: 10.4093/dmj.2014.38.2.150. Epub 2014 Apr 18. PMID 24851209
- [Background] Lingam R, Scott J. Treatment non-adherence in affective disorders. Acta Psychiatr Scand. 2002 Mar;105(3):164-72. doi: 10.1034/j.1600-0447.2002.1r084.x. PMID 11939969
- [Background] Lobo-Escolar A, Roy JF, Saz P, De-la-Camara C, Marcos G, Lobo A; ZARADEMP Workgroup. Association of hypertension with depression in community-dwelling elderly persons: results from the ZARADEMP Project. Psychother Psychosom. 2008;77(5):323-5. doi: 10.1159/000147947. Epub 2008 Jul 25. No abstract available. PMID 18701829
- [Background] Martínez, J.W., Villa Perea, J.A., Jaramillo, J., Quintero, A.M., 2011. Validación del cuestionario de adherencia al tratamiento antihipertensivo Martín Bayarré Grau. Revista Médica de Risaralda, 17(2), 101-105. HTTPS://DOI.ORG/http://dx.doi.org/10.22517/25395203.7595
- [Background] Mann DM, Ponieman D, Leventhal H, Halm EA. Predictors of adherence to diabetes medications: the role of disease and medication beliefs. J Behav Med. 2009 Jun;32(3):278-84. doi: 10.1007/s10865-009-9202-y. Epub 2009 Jan 30. PMID 19184390
- [Background] Martín Alfonso, Libertad, Bayarre Vea, Héctor D, Grau Ábalo, Jorge A., 2008. Validación del cuestionario MBG (Martín-Bayarre-Grau) para evaluar la adherencia terapéutica en hipertensión arterial. Revista Cubana de Salud Pública, 34(1). [citado 2019-08-11]. ISSN 0864-3466. Disponible en: http://scielo.sld.cu/scielo.php?script=sci_arttext&pid=S0864-34662008000100012&lng=es&nrm=iso
- [Background] Markowitz SM, Gonzalez JS, Wilkinson JL, Safren SA. A review of treating depression in diabetes: emerging findings. Psychosomatics. 2011 Jan-Feb;52(1):1-18. doi: 10.1016/j.psym.2010.11.007. PMID 21300190
- [Background] Mezuk B, Eaton WW, Albrecht S, Golden SH. Depression and type 2 diabetes over the lifespan: a meta-analysis. Diabetes Care. 2008 Dec;31(12):2383-90. doi: 10.2337/dc08-0985. PMID 19033418
- [Background] Miller WR, Rollnick S. Motivational interviewing: helping people change. 3rd edn. New York, NY: Guilford Press, 2013.
- [Background] Moliner de la Puente, J.R, Domínguez Sardiña, M, González Paradela, C, Castiñeira Pérez, C, Cespo Sabarís, J.J, Chayan Zas, L, Gonzálvez Rey, J, Pérez García, M, Ríos Rey, M.T, Rodríguez Fernández, M., 2008. Hipertensión arterial in: Guías para la consulta de Atención Primaria. (3a ed.). A Coruña: Casiterides SL.
- [Background] Mullins CD, Whicher D, Reese ES, Tunis S. Generating evidence for comparative effectiveness research using more pragmatic randomized controlled trials. Pharmacoeconomics. 2010;28(10):969-76. doi: 10.2165/11536160-000000000-00000. PMID 20831305
- [Background] Nathan DM. Long-term complications of diabetes mellitus. N Engl J Med. 1993 Jun 10;328(23):1676-85. doi: 10.1056/NEJM199306103282306. No abstract available. PMID 8487827
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Nathan DM, Kuenen J, Borg R, Zheng H, Schoenfeld D, Heine RJ; A1c-Derived Average Glucose Study Group. Translating the A1C assay into estimated average glucose values. Diabetes Care. 2008 Aug;31(8):1473-8. doi: 10.2337/dc08-0545. Epub 2008 Jun 7. PMID 18540046
- [Background] National Clinical Guideline Centre (UK). Hypertension: The Clinical Management of Primary Hypertension in Adults: Update of Clinical Guidelines 18 and 34 [Internet]. London: Royal College of Physicians (UK); 2011 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK83274/ PMID 22855971
- [Background] Nefs G, Pouwer F, Denollet J, Pop V. The course of depressive symptoms in primary care patients with type 2 diabetes: results from the Diabetes, Depression, Type D Personality Zuidoost-Brabant (DiaDDZoB) Study. Diabetologia. 2012 Mar;55(3):608-16. doi: 10.1007/s00125-011-2411-2. Epub 2011 Dec 24. PMID 22198261
- [Background] Nouwen A, Adriaanse MC, van Dam K, Iversen MM, Viechtbauer W, Peyrot M, Caramlau I, Kokoszka A, Kanc K, de Groot M, Nefs G, Pouwer F; European Depression in Diabetes (EDID) Research Consortium. Longitudinal associations between depression and diabetes complications: a systematic review and meta-analysis. Diabet Med. 2019 Dec;36(12):1562-1572. doi: 10.1111/dme.14054. Epub 2019 Jul 31. PMID 31215077
- [Background] Ortiz, M. S., Baeza-Rivera, M. J., & Myers, H. F. (2013). Propiedades psicométricas de la escala de estrés para diabéticos en una muestra de pacientes diabéticos tipo II chilenos. Terapia psicológica, 31(3), 281-286. http://dx.doi.org/10.4067/S0718-48082013000300002
- [Background] O'Shea M, Teeling M, Bennett K. The prevalence and ingredient cost of chronic comorbidity in the Irish elderly population with medication treated type 2 diabetes: a retrospective cross-sectional study using a national pharmacy claims database. BMC Health Serv Res. 2013 Jan 16;13:23. doi: 10.1186/1472-6963-13-23. PMID 23324517
- [Background] Owens-Gary MD, Zhang X, Jawanda S, Bullard KM, Allweiss P, Smith BD. The Importance of Addressing Depression and Diabetes Distress in Adults with Type 2 Diabetes. J Gen Intern Med. 2019 Feb;34(2):320-324. doi: 10.1007/s11606-018-4705-2. Epub 2018 Oct 22. PMID 30350030
- [Background] Patel PJ, Hayward KL, Rudra R, Horsfall LU, Hossain F, Williams S, Johnson T, Brown NN, Saad N, Clouston AD, Stuart KA, Valery PC, Irvine KM, Russell AW, Powell EE. Multimorbidity and polypharmacy in diabetic patients with NAFLD: Implications for disease severity and management. Medicine (Baltimore). 2017 Jun;96(26):e6761. doi: 10.1097/MD.0000000000006761. PMID 28658094
- [Background] Piette JD, Richardson C, Himle J, Duffy S, Torres T, Vogel M, Barber K, Valenstein M. A randomized trial of telephonic counseling plus walking for depressed diabetes patients. Med Care. 2011 Jul;49(7):641-8. doi: 10.1097/MLR.0b013e318215d0c9. PMID 21478777
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Pouwer F, Beekman AT, Nijpels G, Dekker JM, Snoek FJ, Kostense PJ, Heine RJ, Deeg DJ. Rates and risks for co-morbid depression in patients with Type 2 diabetes mellitus: results from a community-based study. Diabetologia. 2003 Jul;46(7):892-8. doi: 10.1007/s00125-003-1124-6. Epub 2003 Jun 18. PMID 12819896
- [Background] Pouwer F, Nefs G, Nouwen A. Adverse effects of depression on glycemic control and health outcomes in people with diabetes: a review. Endocrinol Metab Clin North Am. 2013 Sep;42(3):529-44. doi: 10.1016/j.ecl.2013.05.002. PMID 24011885
- [Background] Powers MA, Bardsley J, Cypress M, Duker P, Funnell MM, Fischl AH, Maryniuk MD, Siminerio L, Vivian E. Diabetes Self-management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. Clin Diabetes. 2016 Apr;34(2):70-80. doi: 10.2337/diaclin.34.2.70. No abstract available. PMID 27092016
- [Background] Renn BN, Feliciano L, Segal DL. The bidirectional relationship of depression and diabetes: a systematic review. Clin Psychol Rev. 2011 Dec;31(8):1239-46. doi: 10.1016/j.cpr.2011.08.001. Epub 2011 Aug 24. PMID 21963669
- [Background] Roy, J. F.; De la Camara, C.; Saz, P.; et al., 2008. Psychosomatic implications in the longitudinal study of late-life depression in the community: The ZARADEMP Project. Journal of Psychosomatic Research, 64(6), 671-671. Web of Science (WOS): 000256455300125
- [Background] Roy, JF; Saz, P; Lobo, A. A longitudinal study of old-age depression in the community: multivariate modelling of psychopathological symptoms to predict incident depression, 2008. Journal of Psychosomatic Research, 59(1), 45-46. Web of Science (WOS): 000232433800096
- [Background] Roy, J. F.; Santabarbara, J.; De-la-Camara, C.; et al, 2010. Cardiovascular burden and long-term risk of first-ever depression: Implications for the vascular depression hypothesis from a population-based study. Journal of Psychosomatic Research, 68(6): 661-661. Web of Science (WOS): 000278468200154
- [Background] Roy T, Lloyd CE, Pouwer F, Holt RI, Sartorius N. Screening tools used for measuring depression among people with Type 1 and Type 2 diabetes: a systematic review. Diabet Med. 2012 Feb;29(2):164-75. doi: 10.1111/j.1464-5491.2011.03401.x. PMID 21824180
- [Background] Santabarbara, J.; Roy, J. F.; De-la-Camara, C.; et al, 2010. History of stroke, incident depressive disorder and competing risk of death. Journal of Psychosomatic Research, 68(6), 662-663. Web of Science (WOS): 000278468200158
- [Background] Safren SA, Gonzalez JS, Wexler DJ, Psaros C, Delahanty LM, Blashill AJ, Margolina AI, Cagliero E. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in patients with uncontrolled type 2 diabetes. Diabetes Care. 2014;37(3):625-33. doi: 10.2337/dc13-0816. Epub 2013 Oct 29. PMID 24170758
- [Background] Saleem T, Mohammad KH, Abdel-Fattah MM, Abbasi AH. Association of glycosylated haemoglobin level and diabetes mellitus duration with the severity of coronary artery disease. Diab Vasc Dis Res. 2008 Sep;5(3):184-9. doi: 10.3132/dvdr.2008.030. PMID 18777491
- [Background] Santos IS, Tavares BF, Munhoz TN, Almeida LS, Silva NT, Tams BD, Patella AM, Matijasevich A. [Sensitivity and specificity of the Patient Health Questionnaire-9 (PHQ-9) among adults from the general population]. Cad Saude Publica. 2013 Aug;29(8):1533-43. doi: 10.1590/0102-311x00144612. Portuguese. PMID 24005919
- [Background] Schechter CB, Cohen HW, Shmukler C, Walker EA. Intervention costs and cost-effectiveness of a successful telephonic intervention to promote diabetes control. Diabetes Care. 2012 Nov;35(11):2156-60. doi: 10.2337/dc12-0048. Epub 2012 Jul 30. PMID 22851599
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Trento M, Raballo M, Trevisan M, Sicuro J, Passera P, Cirio L, Charrier L, Cavallo F, Porta M. A cross-sectional survey of depression, anxiety, and cognitive function in patients with type 2 diabetes. Acta Diabetol. 2012 Jun;49(3):199-203. doi: 10.1007/s00592-011-0275-z. Epub 2011 Mar 27. PMID 21442429
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] van Dam HA, van der Horst FG, Knoops L, Ryckman RM, Crebolder HF, van den Borne BH. Social support in diabetes: a systematic review of controlled intervention studies. Patient Educ Couns. 2005 Oct;59(1):1-12. doi: 10.1016/j.pec.2004.11.001. Epub 2004 Dec 29. PMID 16198213
- [Background] van der Feltz-Cornelis CM, Nuyen J, Stoop C, Chan J, Jacobson AM, Katon W, Snoek F, Sartorius N. Effect of interventions for major depressive disorder and significant depressive symptoms in patients with diabetes mellitus: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):380-95. doi: 10.1016/j.genhosppsych.2010.03.011. Epub 2010 May 15. PMID 20633742
- [Background] van Bastelaar KM, Pouwer F, Geelhoed-Duijvestijn PH, Tack CJ, Bazelmans E, Beekman AT, Heine RJ, Snoek FJ. Diabetes-specific emotional distress mediates the association between depressive symptoms and glycaemic control in Type 1 and Type 2 diabetes. Diabet Med. 2010 Jul;27(7):798-803. doi: 10.1111/j.1464-5491.2010.03025.x. PMID 20636961
- [Background] Verma SK, Luo N, Subramaniam M, Sum CF, Stahl D, Liow PH, Chong SA. Impact of depression on health related quality of life in patients with diabetes. Ann Acad Med Singap. 2010 Dec;39(12):913-7. PMID 21274488
- [Background] Vermeire E, Wens J, Van Royen P, Biot Y, Hearnshaw H, Lindenmeyer A. Interventions for improving adherence to treatment recommendations in people with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2005 Apr 18;2005(2):CD003638. doi: 10.1002/14651858.CD003638.pub2. PMID 15846672
- [Background] Vink NM, Klungel OH, Stolk RP, Denig P. Comparison of various measures for assessing medication refill adherence using prescription data. Pharmacoepidemiol Drug Saf. 2009 Feb;18(2):159-65. doi: 10.1002/pds.1698. PMID 19109809
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Background] World Health Organization, 2019. Body Mass Index. Extracted from: http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthy-lifestyle/body-mass-index-bmi
- [Background] Yasmin F, Banu B, Zakir SM, Sauerborn R, Ali L, Souares A. Positive influence of short message service and voice call interventions on adherence and health outcomes in case of chronic disease care: a systematic review. BMC Med Inform Decis Mak. 2016 Apr 22;16:46. doi: 10.1186/s12911-016-0286-3. PMID 27106263
- [Derived] Gomez-Barrera M, Lozano-Del Hoyo ML, Roy JF, Fernandez-Rodrigo MT, Gomez-Torres P, Blazquez-Ornat I, Perez-Calahorra S, Samaniego Diaz de Corcuera ME, Ferrer-Lopez E, Ramon-Arbues E. Nurse-Led Telephone Program for Nonadherent to Treatment Type 2 Diabetics With Comorbid Depression: A Cost-Consequence and Budget Impact Analysis. J Nurs Manag. 2024 Nov 20;2024:9989080. doi: 10.1155/2024/9989080. eCollection 2024. PMID 40224867